CLINICAL TRIAL: NCT02638493
Title: IGHID 11526 - The Compartmental Biology of HIV in the Male Genital Tract
Brief Title: The Compartmental Biology of HIV in the Male Genital Tract
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Julie Dumond, PharmD, Assistant Professor, University of North Carolina, Chapel Hill
Other Study IDs: 15-2767; R01DK108424-01 (NIH)
Record Dates: First submitted 2015-12-10; First posted 2015-12-23 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-04

CONDITIONS: Human Immunodeficiency Virus; Virus Shedding
Keywords: HIV; tenofovir-emtricitabine; antiretroviral therapy; Prevention; tenofovir alafenamide
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and semen samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV positive TDF/FTC: 8 HIV positive men taking TDF/FTC as treatment
- HIV negative: 8 HIV negative men taking TDF/FTC as pre-exposure prophylaxis
- HIV Positive TAF: 8 HIV positive men taking TAF as treatment

SUMMARY:
Male participants taking tenofovir-emtricitabine (TDF/FTC) will provide semen and blood samples which will be analyzed to better understand the pharmacology of antiretroviral therapy in the male genital tract.

DETAILED DESCRIPTION:
8 HIV positive men taking TDF/FTC and 8 HIV negative men taking TDF/FTC as pre-exposure prophylaxis will provide multiple semen and blood samples during a 48-hour inpatient visit. 8 HIV positive men taking TAF (tenofovir alafenamide) will provide multiple semen and blood samples during a 48-hour inpatient visit.

Participants will take part in the study for approximately two months. After the screening visit, there is one 2 day overnight visit for intensive PK/PD (pharmacokinetic/pharmacodynamic) sampling. The investigators will study drug concentrations and intracellular endogenous nucleotide concentrations (dATP and dCTP) in seminal plasma and (where appropriate) seminal cells.

Samples will be analyzed through the use of novel laboratory methods to determine the seminal plasma and seminal cell concentrations of tenofovir and emtricitabine. New technologies will be used to better understand compartmental and intracellular antiretroviral pharmacology of nucleoside/tide reverse transcriptase inhibitors. Pharmacokinetic modeling will be used to estimate the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Born male between the ages of 18 and 60
* HIV positive taking TDF/FTC (and a third drug) as treatment; or HIV negative men receiving TDF/FTC as pre-exposure prophylaxis; HIV positive men taking tenofovir alafenamide
* if on routine treatment must have been taking medication for at least 3 months and adherence to medication as assessed by blood plasma HIV RNA less than 50 copies per mL.
* documentation of at least 80% adherence to antiretroviral (ART) regimen, through clinician or self-report, with no missed doses in the 3 days prior to the inpatient visit.
* willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurologic disease that would pose unnecessary risk or interfere with study results.
* unwilling or unable to abstain from sexual activity 72 hours prior to overnight sampling visit
* unlikely to remain on current drug regimen during study period
* anemia that precludes blood donation
* unable to provide semen specimen
* current receipt of other medications that may affect endogenous nucleotide concentrations, such as additional HIV nucleoside reverse transcriptase inhibitors, ribavirin, or adefovir

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: HIV positive and HIV negative men taking TDF/FTC once daily, HIV positive men taking TAF/FTC once daily
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Dumond, PharmD, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galvin SR, Cohen MS. The role of sexually transmitted diseases in HIV transmission. Nat Rev Microbiol. 2004 Jan;2(1):33-42. doi: 10.1038/nrmicro794. PMID 15035007
- [Background] Cohen MS, Gay C, Kashuba AD, Blower S, Paxton L. Narrative review: antiretroviral therapy to prevent the sexual transmission of HIV-1. Ann Intern Med. 2007 Apr 17;146(8):591-601. doi: 10.7326/0003-4819-146-8-200704170-00010. PMID 17438318
- [Background] Anderson DJ, Politch JA, Nadolski AM, Blaskewicz CD, Pudney J, Mayer KH. Targeting Trojan Horse leukocytes for HIV prevention. AIDS. 2010 Jan 16;24(2):163-87. doi: 10.1097/QAD.0b013e32833424c8. No abstract available. PMID 20010071
- [Background] Joseph SB, Swanstrom R, Kashuba AD, Cohen MS. Bottlenecks in HIV-1 transmission: insights from the study of founder viruses. Nat Rev Microbiol. 2015 Jul;13(7):414-25. doi: 10.1038/nrmicro3471. Epub 2015 Jun 8. PMID 26052661
- See also: University of North Carolina website — http://www.unc.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at the University of North Carolina at Chapel Hill and surrounding areas, through Institutional Review Board (IRB)-approved advertisements.
Pre-assignment Details: Participants interested in the study were pre-screened for eligibility using an IRB-approved questionnaire.
Groups:
- HIV Positive TDF/FTC: 8 HIV positive men taking TDF/FTC (Tenofovir Disoproxil Fumarate/Emtricitabine) as treatment
- HIV Negative: 8 HIV negative men taking TDF/FTC (Tenofovir Disoproxil Fumarate/Emtricitabine) as pre-exposure prophylaxis
- HIV Positive TAF: 8 HIV positive men taking TAF (Tenofovir Alafenamide) as treatment
Period: Overall Study
Arm/Group | HIV Positive TDF/FTC | HIV Negative | HIV Positive TAF
Started | 10 (Two men were not able to provide semen samples, and thus were replaced) | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 2 | 0 | 0
Not completed — Inability to provide semen samples | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Positive TDF/FTC | HIV Negative | HIV Positive TAF | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 36.5 [33 to 41] | 30.5 [19 to 39] | 45.5 [34 to 52] | 36.5 [19 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 8 | 8 | 24
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Semen Clearance (CL) of Tenofovir
Description: Samples will be analyzed for drug concentrations at the following time points post dose: 3, 6, 9, 12, 18 and 24 hours, and used to estimate clearance from semen from a 300mg dose of tenofovir.
Time Frame: Samples collected at 3, 6, 9, 12, 18 and 24 hours post-dose
Measure: Median (Inter-Quartile Range); unit: L/hr
Arm/Group | HIV Positive TDF/FTC | HIV Negative | HIV Positive TAF
Number analyzed (Participants) | 8 | 8 | 8
L/hr | 33.88 [18.86 to 65.26] | 51.21 [19.18 to 77.79] | 5.65 [3.23 to 7.23]

2. Primary Outcome: Semen Clearance (CL) of Emtricitabine
Description: Samples will be analyzed for drug concentration at the following time points post dose: 3, 6, 9, 12, 18 and 24 hours, and used to estimate clearance from semen from a 200mg dose of emtricitabine.
Time Frame: Samples collected at 3, 6, 9, 12, 18 and 24 hours post-dose
Measure: Median (Inter-Quartile Range); unit: L/hr
Arm/Group | HIV Positive TDF/FTC | HIV Negative | HIV Positive TAF
Number analyzed (Participants) | 8 | 8 | 8
L/hr | 5.91 [5.43 to 8.28] | 8.72 [4.95 to 12.30] | 7.12 [3.91 to 11.09]

3. Primary Outcome: Semen Clearance (CL) of Tenofovir Diphosphate
Description: Samples will be analyzed for drug concentration at the following time points post dose: 3, 6, 9, 12, 18 and 24 hours, and used to estimate the clearance of tenofovir diphosphate, an intracellular metabolite of tenofovir, from seminal mononuclear cells, following a 300mg dose of tenofovir.
Time Frame: Samples collected at 3, 6, 9, 12, 18 and 24 hours post-dose
Measure: Median (Inter-Quartile Range); unit: fmol/10x6 cells
Arm/Group | HIV Positive TDF/FTC | HIV Negative | HIV Positive TAF
Number analyzed (Participants) | 8 | 8 | 8
fmol/10x6 cells | 21 [5.7 to 88] | 21 [4.2 to 91] | 35 [24 to 78]

4. Primary Outcome: Semen Clearance (CL) of Emtricitabine Triphosphate
Description: Samples will be analyzed for drug concentration at the following time points post dose: 3, 6, 9, 12, 18 and 24 hours, and used to estimate the clearance of emtricitabine triphosphate, an intracellular metabolite of emtricitabine, from seminal mononuclear cells, following a 200mg dose of emtricitabine.
Time Frame: Samples collected at 3, 6, 9, 12, 18 and 24 hours post-dose
Population: Semen (SMC) Steady State Concentrations (Css,ave) of Emtricitabine Triphosphate
Measure: Median (Inter-Quartile Range); unit: fmol/10 E6 cells
Arm/Group | HIV Positive TDF/FTC | HIV Negative | HIV Positive TAF
Number analyzed (Participants) | 8 | 8 | 8
fmol/10 E6 cells | 59 [22 to 119] | 90 [34 to 193] | 179 [108 to 395]

5. Primary Outcome: Peripheral Blood Mononuclear Cell (PBMC) Clearance (CL) of Tenofovir Diphosphate
Description: Samples will be analyzed for drug concentration at the following time points post dose: 3, 6, 9, 12, 18 and 24 hours, and used to estimate the clearance of tenofovir diphosphate, an intracellular metabolite of tenofovir, from peripheral blood mononuclear cells, following a 300mg dose of tenofovir.
Time Frame: Samples collected at 3, 6, 9, 12, 18 and 24 hours post-dose
Measure: Median (Inter-Quartile Range); unit: fmol/10 E6 cells
Arm/Group | HIV Positive TDF/FTC | HIV Negative | HIV Positive TAF
Number analyzed (Participants) | 8 | 8 | 8
fmol/10 E6 cells | 174 [115 to 239] | 119 [76 to 174] | 935 [684 to 2024]

6. Primary Outcome: Peripheral Blood Mononuclear Cell (PBMC) Clearance (CL) of Emtricitabine Triphosphate
Description: Samples will be analyzed for drug concentration at the following time points post dose: 3, 6, 9, 12, 18 and 24 hours, and used to estimate the clearance of emtricitabine triphosphate, an intracellular metabolite of emtricitabine, from peripheral blood mononuclear cells, following a 200mg dose of emtricitabine.
Time Frame: Samples collected at 3, 6, 9, 12, 18 and 24 hours post-dose
Measure: Median (Inter-Quartile Range); unit: fmol/10 E6 cells
Arm/Group | HIV Positive TDF/FTC | HIV Negative | HIV Positive TAF
Number analyzed (Participants) | 8 | 8 | 8
fmol/10 E6 cells | 6038 [4465 to 10088] | 6135 [3889 to 8303] | 8242 [5602 to 13480]

7. Secondary Outcome: Tenofovir Diphosphate (TFVdp)/Deoxyadenosine Triphosphate (dATP) Ratio in Seminal Mononuclear Cells
Description: dATP concentrations in seminal mononuclear cells will be measured and compared to tenofovir diphosphate concentrations, using a ratio, and summarized descriptively for each subject, as well as across subjects. As the six seminal cell samples collected per man were pooled for analysis due to low cell recovery, a single ratio value per participant was calculated and summarized by study arm.
Time Frame: Average concentration in a 24 hour dosing interval
Measure: Median (Inter-Quartile Range); unit: TFVdp:dATP ratio
Arm/Group | HIV Positive TDF/FTC | HIV Negative | HIV Positive TAF
Number analyzed (Participants) | 8 | 8 | 8
TFVdp:dATP ratio | 0.99 [0.43 to 1.54] | 0.66 [0.22 to 1.21] | 1.10 [0.42 to 1.70]

8. Secondary Outcome: Emtricitabine Triphosphate (FTCtp)/Deoxyadenosine Triphosphate (dCTP) Ratio in Seminal Mononuclear Cells
Description: dCTP concentrations in seminal mononuclear cells will be measured and compared to emtricitabine triphosphate concentrations, using a ratio, and summarized descriptively for each subject, as well as across subjects. As the six seminal cell samples collected per man were pooled for analysis due to low cell recovery, a single ratio value per participant was calculated and summarized by study arm.
Time Frame: Average concentration in a 24 hour dosing interval
Measure: Median (Inter-Quartile Range); unit: FTCtp:dCTP ratio
Arm/Group | HIV Positive TDF/FTC | HIV Negative | HIV Positive TAF
Number analyzed (Participants) | 8 | 8 | 8
FTCtp:dCTP ratio | 0.52 [0.38 to 1.14] | 0.96 [0.39 to 1.85] | 3.81 [2.30 to 3.98]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent, until end of study enrollment.
Description: does not differ
Arm/Group | HIV Positive TDF/FTC | HIV Negative | HIV Positive TAF
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 1/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV Positive TDF/FTC (N=8) | HIV Negative (N=8) | HIV Positive TAF (N=8)
Viral Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Sore throat and temperature reported, rapid strep sent, result negative.
Penile skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Mild skin irritation/soreness following sample

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes